CLINICAL TRIAL: NCT01032356
Title: Contracture Reduction Following Distal Radius Fracture Surgical Management
Brief Title: Dynasplint for Distal Radius Fracture
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Dynasplint Systems, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: WED1
Record Dates: First submitted 2009-12-11; First posted 2009-12-15 (Estimated); Last update posted 2013-07-11 (Estimated); Status verified 2013-07

CONDITIONS: Distal Radius Fracture
Keywords: Distal Radius fracture
MeSH Terms: conditions — Wrist Fractures

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Dynasplint (Experimental): Patients will be treated with the current standard of care and the Wrist Extension Dynasplint.
  Interventions: Device: Wrist Extension Dynasplint

INTERVENTIONS:
Device: Wrist Extension Dynasplint — Dynamic splinting utilizes the protocols of Low-Load Prolonged Stretch (LLPS) with calibrated adjustable tension to increase Total End Range Time (TERT)to reduce contracture. The Dynasplint or "Experimental" group will add this therapy to their standard of care regimen

SUMMARY:
The purpose of this study was to examine the efficacy of dynamic splinting as a therapeutic modality in reducing contracture following surgical treatment of distal radius fractures.

ELIGIBILITY:
Inclusion Criteria:

* Distal radius fracture treated with surgical management and wrist flexion contracture upon follow up

Exclusion Criteria:

* Carpal Fractures (Scaphoid, Lunate, Hamate, and Trapezium)
* Radial nerve entrapment
* Arthrodesis
* Traumatic dislocation of the distal ulna

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Estimated)
Dates: Start 2016-01; Primary Completion 2016-06 (Estimated)

PRIMARY OUTCOMES:
The dependent variable will be change in maximal, active range of motion in extension and the independent variables will include DASH scores and measurements taken from radiographic imaging | 12 weeks

REFERENCES:
- [Background] 1) Berner SH, Willis FB. Treatment of Carpal Tunnel Syndrome with Dynasplint: a Randomized, Controlled Trial. Journal of Medicine, 2008 Dec 1(1), pg 90-94
- [Background] Fanuele J, Koval KJ, Lurie J, Zhou W, Tosteson A, Ring D. Distal radial fracture treatment: what you get may depend on your age and address. J Bone Joint Surg Am. 2009 Jun;91(6):1313-9. doi: 10.2106/JBJS.H.00448. PMID 19487507
- [Background] Franko OI, Zurakowski D, Day CS. Functional disability of the wrist: direct correlation with decreased wrist motion. J Hand Surg Am. 2008 Apr;33(4):485-92. doi: 10.1016/j.jhsa.2008.01.005. PMID 18406951
- [Background] Handoll HH, Huntley JS, Madhok R. Different methods of external fixation for treating distal radial fractures in adults. Cochrane Database Syst Rev. 2008 Jan 23;2008(1):CD006522. doi: 10.1002/14651858.CD006522.pub2. PMID 18254105
- [Background] Lai JM, Francisco GE, Willis FB. Dynamic splinting after treatment with botulinum toxin type-A: a randomized controlled pilot study. Adv Ther. 2009 Feb;26(2):241-8. doi: 10.1007/s12325-008-0139-2. Epub 2009 Feb 4. PMID 19194671
- [Background] Lutz M, Rudisch A, Kralinger F, Smekal V, Goebel G, Gabl M, Pechlaner S. Sagittal wrist motion of carpal bones following intraarticular fractures of the distal radius. J Hand Surg Br. 2005 Jun;30(3):282-7. doi: 10.1016/j.jhsb.2004.12.012. Epub 2005 Apr 8. PMID 15862369
- [Background] Maciel JS, Taylor NF, McIlveen C. A randomised clinical trial of activity-focussed physiotherapy on patients with distal radius fractures. Arch Orthop Trauma Surg. 2005 Oct;125(8):515-20. doi: 10.1007/s00402-005-0037-x. Epub 2005 Oct 22. PMID 16136342
- [Background] McKee P, Nguyen C. Customized dynamic splinting: orthoses that promote optimal function and recovery after radial nerve injury: a case report. J Hand Ther. 2007 Jan-Mar;20(1):73-87; quiz 88. doi: 10.1197/j.jht.2006.11.013. PMID 17254911
- [Background] Nagy L. Salvage of post-traumatic arthritis following distal radius fracture. Hand Clin. 2005 Aug;21(3):489-98. doi: 10.1016/j.hcl.2005.03.005. PMID 16039459
- [Background] Saini R, Gill SS, Dhillon MS, Goyal T, Wardak E, Prasad P. Results of dorsal approach in surgical correction of congenital vertical talus: an Indian experience. J Pediatr Orthop B. 2009 Mar;18(2):63-8. doi: 10.1097/BPB.0b013e328321ce71. PMID 19106803
- [Background] Shin EK, Jupiter JB. Current concepts in the management of distal radius fractures. Acta Chir Orthop Traumatol Cech. 2007 Aug;74(4):233-46. PMID 17877939
- [Background] Watt CF, Taylor NF, Baskus K. Do Colles' fracture patients benefit from routine referral to physiotherapy following cast removal? Arch Orthop Trauma Surg. 2000;120(7-8):413-5. doi: 10.1007/pl00013772. PMID 10968529
- [Background] Wilcke MK, Abbaszadegan H, Adolphson PY. Patient-perceived outcome after displaced distal radius fractures. A comparison between radiological parameters, objective physical variables, and the DASH score. J Hand Ther. 2007 Oct-Dec;20(4):290-8; quiz 299. doi: 10.1197/j.jht.2007.06.001. PMID 17954350
- [Background] Willis B, Gaspar P, Neffendorf C. Device and Physical Therapy to Unfreeze Shoulder Motion. BioMechanics. 2007 Jan:14(1):45-49